CLINICAL TRIAL: NCT02758288
Title: BK Viremia and BK Virus Nephropathy Post Kidney Transplant Comparison of New Practices With Traditional Approach: A Combined Retrospective Chart Review and Prospective Observational Study
Brief Title: BK Virus Post-Kidney Transplant: New Practice Versus Traditional Approach
Status: Withdrawn | Type: Observational
Sponsor: Loma Linda University (Other)
Responsible Party: Principal Investigator, Amir Abdipour, MD, Assistant Professor of Medicine, Loma Linda University
Other Study IDs: 5150278
Record Dates: First submitted 2016-03-02; First posted 2016-05-02 (Estimated); Last update posted 2020-10-05 (Actual); Status verified 2020-10

CONDITIONS: BK Virus Infection; BK Virus Nephropathy
Keywords: Kidney transplant; BK Viremia; BK Nephropathy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- New Protocol to treat BK viremia or BKVAN: Adult kidney recipients who are determined to have BK viremia with a BK PCR viral load over 500 copy post-transplant treated with a new treatment protocol, prospective data collection approach
  Interventions: Other: New Protocol - BK viremia or BK virus nephropathy
- Standard Protocol to treat BK viremia or BKVAN: Adult kidney recipients who are determined to have BK viremia with a BK PCR viral load over 500 copy post-transplant treated with a traditional standard of care protocol, retrospective data collection approach
  Interventions: Other: Standard Protocol - BK viremia or BK virus nephropathy

INTERVENTIONS:
Other: New Protocol - BK viremia or BK virus nephropathy — Data collected prospectively that will follow new clinical practice guidelines that were developed by Loma Linda Nephrology group with collaboration with Transplant surgeons to improve care of patients complicated with BK viremia or BK virus nephropathy.
  Groups: New Protocol to treat BK viremia or BKVAN
Other: Standard Protocol - BK viremia or BK virus nephropathy — Data collected retrospectively that followed standard clinical practice guidelines that were developed by Loma Linda Nephrology group with collaboration with Transplant surgeons to improve care of patients complicated with BK viremia or BK virus nephropathy.
  Groups: Standard Protocol to treat BK viremia or BKVAN

SUMMARY:
The investigator's aim in this study is to evaluate the impact of a new standard of care protocol for the treatment of BK viremia and nephropathy (BKVAN), which includes switching from Tacrolimus to equivalent dose of Cyclosporine in patients who have been diagnosed with BK viremia or BKVAN based on their viral load, overall graft function (estimated glomerular filtration rate), acute rejection, and rate of graft loss due to rejection or BKVAN.

DETAILED DESCRIPTION:
This study will be a combined retrospective chart review and prospective observational study. This will be a single center project that will take place at Loma Linda University Transplant Institute. All adult kidney recipients who are determined to have BK viremia with a BK PCR viral load over 500 copy post-transplant and meet the inclusion criteria but no exclusion criteria will be enrolled and observed per study protocol.

All kidney transplant recipients are routinely assessed for BK virus nephropathy and viremia post transplant as part of their standard care. Patients with BK viremia or BK virus nephropathy will have adjustments in their immunosuppressive medication based on current guidelines and recommendations which include reduction in immunosuppression, treatment with medications with antiviral activity (Cidofovir, Ciprofloxacin, Leflunomide, IVIG) or switching from a Tacrolimus (Prograf)-based regimen to a Cyclosporine-based regimen. Retrospectively, the investigator will collect data on patients who have been diagnosed with BK viremia or BK virus nephropathy and have had such a management in past 66 months (from 1/1/2010 till 06/30/2015). Prospectively, the investigator will enroll and collect data on patients who will be treated for BK viremia or BK virus nephropathy.

As standard of care, all kidney transplant recipients will be seen routinely on weekly-biweekly basis in post-transplant clinic for up to 3 months then every 3 months for up to a year and yearly thereafter. All kidney transplant recipients will be monitored for BK viremia by having blood PCR tested on a monthly basis at 1, 2, 3, 6, and 12 months after transplant. Also, all patients post-kidney transplant will be tested for BK viremia if there is an acute rise in their creatinine.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Recipient of kidney or combined kidney and pancreas

  * BK viremia confirmed with blood PCR test with viral load over 500
  * BK virus nephropathy confirmed by kidney biopsy

Exclusion Criteria:

* Recipient of combined organ transplant except kidney and pancreases
* Patient age < 18 years
* If patient does not consent for kidney biopsy
* Currently on treatment for acute rejection
* Patients with HIV, Hep C or Hep B infection
* Patients who are on other immunosuppression beside our standard regimen which includes Prograf, cellcept / Myfortic and prednisone

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult kidney recipients who are determined to have BK viremia post-transplant
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2015-09; Primary Completion 2021-07 (Estimated); Study Completion 2022-07 (Estimated)

PRIMARY OUTCOMES:
Kidney function to compare effectiveness of a new care protocol for the treatment of BK viremia (BK PCR viral load over 500 copy) and BKVAN (confirmed by kidney biopsy) with a similar cohort treated with traditional methods. | 12 months

SECONDARY OUTCOMES:
Rate of BK nephropathy in both treatment groups confirmed by kidney biopsy | 24 months
Rate of acute cellular or humoral rejection in both treatment groups confirmed by kidney biopsy | 24 months
Rate of graft loss in both group as determined by elevated creatinine level and kidney biopsy | 24 months
Estimated glomerular filtration rate (eGFR) at start of the study (0) , 3, 6, 12 and 24 months between two groups | 3, 6, 12, 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Amir Abdipour, MD, Principal Investigator — Loma Linda University Health
Locations (1):
- Loma Linda University Medical Center, Loma Linda, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tonelli M, Wiebe N, Knoll G, Bello A, Browne S, Jadhav D, Klarenbach S, Gill J. Systematic review: kidney transplantation compared with dialysis in clinically relevant outcomes. Am J Transplant. 2011 Oct;11(10):2093-109. doi: 10.1111/j.1600-6143.2011.03686.x. Epub 2011 Aug 30. PMID 21883901
- [Background] Port FK, Wolfe RA, Mauger EA, Berling DP, Jiang K. Comparison of survival probabilities for dialysis patients vs cadaveric renal transplant recipients. JAMA. 1993 Sep 15;270(11):1339-43. PMID 8360969
- [Background] Schnuelle P, Lorenz D, Trede M, Van Der Woude FJ. Impact of renal cadaveric transplantation on survival in end-stage renal failure: evidence for reduced mortality risk compared with hemodialysis during long-term follow-up. J Am Soc Nephrol. 1998 Nov;9(11):2135-41. doi: 10.1681/ASN.V9112135. PMID 9808102
- [Background] Padgett BL, Walker DL. Prevalence of antibodies in human sera against JC virus, an isolate from a case of progressive multifocal leukoencephalopathy. J Infect Dis. 1973 Apr;127(4):467-70. doi: 10.1093/infdis/127.4.467. No abstract available. PMID 4571704
- [Background] Bressollette-Bodin C, Coste-Burel M, Hourmant M, Sebille V, Andre-Garnier E, Imbert-Marcille BM. A prospective longitudinal study of BK virus infection in 104 renal transplant recipients. Am J Transplant. 2005 Aug;5(8):1926-33. doi: 10.1111/j.1600-6143.2005.00934.x. PMID 15996241
- [Background] Ginevri F, Azzi A, Hirsch HH, Basso S, Fontana I, Cioni M, Bodaghi S, Salotti V, Rinieri A, Botti G, Perfumo F, Locatelli F, Comoli P. Prospective monitoring of polyomavirus BK replication and impact of pre-emptive intervention in pediatric kidney recipients. Am J Transplant. 2007 Dec;7(12):2727-35. doi: 10.1111/j.1600-6143.2007.01984.x. Epub 2007 Oct 1. PMID 17908275
- [Background] Brennan DC, Agha I, Bohl DL, Schnitzler MA, Hardinger KL, Lockwood M, Torrence S, Schuessler R, Roby T, Gaudreault-Keener M, Storch GA. Incidence of BK with tacrolimus versus cyclosporine and impact of preemptive immunosuppression reduction. Am J Transplant. 2005 Mar;5(3):582-94. doi: 10.1111/j.1600-6143.2005.00742.x. PMID 15707414
- [Background] Kadambi PV, Josephson MA, Williams J, Corey L, Jerome KR, Meehan SM, Limaye AP. Treatment of refractory BK virus-associated nephropathy with cidofovir. Am J Transplant. 2003 Feb;3(2):186-91. doi: 10.1034/j.1600-6143.2003.30202.x. PMID 12614296
- [Background] Moscarelli L, Caroti L, Antognoli G, Zanazzi M, Di Maria L, Carta P, Minetti E. Everolimus leads to a lower risk of BKV viremia than mycophenolic acid in de novo renal transplantation patients: a single-center experience. Clin Transplant. 2013 Jul-Aug;27(4):546-54. doi: 10.1111/ctr.12151. Epub 2013 Jun 13. PMID 23758330
- [Background] Araya CE, Garin EH, Neiberger RE, Dharnidharka VR. Leflunomide therapy for BK virus allograft nephropathy in pediatric and young adult kidney transplant recipients. Pediatr Transplant. 2010 Feb;14(1):145-50. doi: 10.1111/j.1399-3046.2009.01183.x. Epub 2009 Mar 31. PMID 19344337
- [Background] Williams JW, Javaid B, Kadambi PV, Gillen D, Harland R, Thistlewaite JR, Garfinkel M, Foster P, Atwood W, Millis JM, Meehan SM, Josephson MA. Leflunomide for polyomavirus type BK nephropathy. N Engl J Med. 2005 Mar 17;352(11):1157-8. doi: 10.1056/NEJM200503173521125. No abstract available. PMID 15784677
- [Background] Leung AY, Chan MT, Yuen KY, Cheng VC, Chan KH, Wong CL, Liang R, Lie AK, Kwong YL. Ciprofloxacin decreased polyoma BK virus load in patients who underwent allogeneic hematopoietic stem cell transplantation. Clin Infect Dis. 2005 Feb 15;40(4):528-37. doi: 10.1086/427291. Epub 2005 Jan 21. PMID 15712075
- [Background] Randhawa PS. Anti-BK virus activity of ciprofloxacin and related antibiotics. Clin Infect Dis. 2005 Nov 1;41(9):1366-7; author reply 1367. doi: 10.1086/497080. No abstract available. PMID 16206122
- [Background] Hirsch HH, Vincenti F, Friman S, Tuncer M, Citterio F, Wiecek A, Scheuermann EH, Klinger M, Russ G, Pescovitz MD, Prestele H. Polyomavirus BK replication in de novo kidney transplant patients receiving tacrolimus or cyclosporine: a prospective, randomized, multicenter study. Am J Transplant. 2013 Jan;13(1):136-45. doi: 10.1111/j.1600-6143.2012.04320.x. Epub 2012 Nov 8. PMID 23137180
- [Background] Renner FC, Dietrich H, Bulut N, Celik D, Freitag E, Gaertner N, Karoui S, Mark J, Raatz C, Weimer R, Feustel A. The risk of polyomavirus-associated graft nephropathy is increased by a combined suppression of CD8 and CD4 cell-dependent immune effects. Transplant Proc. 2013 May;45(4):1608-10. doi: 10.1016/j.transproceed.2013.01.026. PMID 23726630
- [Background] Huang G, Chen LZ, Qiu J, Wang CX, Fei JG, Deng SX, Li J, Chen GD, Zhang L, Fu Q, Zeng WT, Zhao DQ. Prospective study of polyomavirus BK replication and nephropathy in renal transplant recipients in China: a single-center analysis of incidence, reduction in immunosuppression and clinical course. Clin Transplant. 2010 Sep-Oct;24(5):599-609. doi: 10.1111/j.1399-0012.2009.01141.x. PMID 19925472
- [Background] Knoll GA, Bell RC. Tacrolimus versus cyclosporin for immunosuppression in renal transplantation: meta-analysis of randomised trials. BMJ. 1999 Apr 24;318(7191):1104-7. doi: 10.1136/bmj.318.7191.1104. PMID 10213717
- [Background] Alghamdi S, Nabi Z, Skolnik E, Alkorbi L, Albaqumi M. Cyclosporine versus tacrolimus maintenance therapy in renal transplant. Exp Clin Transplant. 2011 Jun;9(3):170-4. PMID 21649564
- [Background] Gardner SD, Field AM, Coleman DV, Hulme B. New human papovavirus (B.K.) isolated from urine after renal transplantation. Lancet. 1971 Jun 19;1(7712):1253-7. doi: 10.1016/s0140-6736(71)91776-4. No abstract available. PMID 4104714
- [Background] Boothpur R, Brennan DC. Human polyoma viruses and disease with emphasis on clinical BK and JC. J Clin Virol. 2010 Apr;47(4):306-12. doi: 10.1016/j.jcv.2009.12.006. Epub 2010 Jan 8. PMID 20060360
- [Background] Elphick GF, Querbes W, Jordan JA, Gee GV, Eash S, Manley K, Dugan A, Stanifer M, Bhatnagar A, Kroeze WK, Roth BL, Atwood WJ. The human polyomavirus, JCV, uses serotonin receptors to infect cells. Science. 2004 Nov 19;306(5700):1380-3. doi: 10.1126/science.1103492. PMID 15550673
- [Background] Monaco MC, Jensen PN, Hou J, Durham LC, Major EO. Detection of JC virus DNA in human tonsil tissue: evidence for site of initial viral infection. J Virol. 1998 Dec;72(12):9918-23. doi: 10.1128/JVI.72.12.9918-9923.1998. PMID 9811728
- [Background] Rinaldo CH, Tylden GD, Sharma BN. The human polyomavirus BK (BKPyV): virological background and clinical implications. APMIS. 2013 Aug;121(8):728-45. doi: 10.1111/apm.12134. Epub 2013 Jun 19. PMID 23782063
- [Background] Balba GP, Javaid B, Timpone JG Jr. BK polyomavirus infection in the renal transplant recipient. Infect Dis Clin North Am. 2013 Jun;27(2):271-83. doi: 10.1016/j.idc.2013.02.002. Epub 2013 Apr 17. PMID 23714340
- [Background] Nickeleit V, Klimkait T, Binet IF, Dalquen P, Del Zenero V, Thiel G, Mihatsch MJ, Hirsch HH. Testing for polyomavirus type BK DNA in plasma to identify renal-allograft recipients with viral nephropathy. N Engl J Med. 2000 May 4;342(18):1309-15. doi: 10.1056/NEJM200005043421802. PMID 10793163
- [Background] Vasudev B, Hariharan S, Hussain SA, Zhu YR, Bresnahan BA, Cohen EP. BK virus nephritis: risk factors, timing, and outcome in renal transplant recipients. Kidney Int. 2005 Oct;68(4):1834-9. doi: 10.1111/j.1523-1755.2005.00602.x. PMID 16164661
- [Background] Randhawa P, Ho A, Shapiro R, Vats A, Swalsky P, Finkelstein S, Uhrmacher J, Weck K. Correlates of quantitative measurement of BK polyomavirus (BKV) DNA with clinical course of BKV infection in renal transplant patients. J Clin Microbiol. 2004 Mar;42(3):1176-80. doi: 10.1128/JCM.42.3.1176-1180.2004. PMID 15004071
- [Background] Kahan AV, Coleman DV, Koss LG. Activation of human polyomavirus infection-detection by cytologic technics. Am J Clin Pathol. 1980 Sep;74(3):326-32. doi: 10.1093/ajcp/74.3.326. PMID 6251715
- [Background] Hirsch HH, Randhawa P; AST Infectious Diseases Community of Practice. BK virus in solid organ transplant recipients. Am J Transplant. 2009 Dec;9 Suppl 4:S136-46. doi: 10.1111/j.1600-6143.2009.02904.x. No abstract available. PMID 20070673
- [Background] Hariharan S. BK virus nephritis after renal transplantation. Kidney Int. 2006 Feb;69(4):655-62. doi: 10.1038/sj.ki.5000040. PMID 16395271
- [Background] Drachenberg CB, Hirsch HH, Ramos E, Papadimitriou JC. Polyomavirus disease in renal transplantation: review of pathological findings and diagnostic methods. Hum Pathol. 2005 Dec;36(12):1245-55. doi: 10.1016/j.humpath.2005.08.009. Epub 2005 Oct 19. PMID 16311117
- [Background] Hirsch HH, Steiger J. Polyomavirus BK. Lancet Infect Dis. 2003 Oct;3(10):611-23. doi: 10.1016/s1473-3099(03)00770-9. PMID 14522260
- [Background] Binet I, Nickeleit V, Hirsch HH, Prince O, Dalquen P, Gudat F, Mihatsch MJ, Thiel G. Polyomavirus disease under new immunosuppressive drugs: a cause of renal graft dysfunction and graft loss. Transplantation. 1999 Mar 27;67(6):918-22. doi: 10.1097/00007890-199903270-00022. PMID 10199744
- [Background] Ramos E, Drachenberg CB, Papadimitriou JC, Hamze O, Fink JC, Klassen DK, Drachenberg RC, Wiland A, Wali R, Cangro CB, Schweitzer E, Bartlett ST, Weir MR. Clinical course of polyoma virus nephropathy in 67 renal transplant patients. J Am Soc Nephrol. 2002 Aug;13(8):2145-51. doi: 10.1097/01.asn.0000023435.07320.81. PMID 12138148
- [Background] Ronco C. Biomarkers for acute kidney injury: is NGAL ready for clinical use? Crit Care. 2014 Dec 10;18(6):680. doi: 10.1186/s13054-014-0680-0. PMID 25672254
- [Background] Han SB, Cho B, Kang JH. BK virus-associated hemorrhagic cystitis after pediatric stem cell transplantation. Korean J Pediatr. 2014 Dec;57(12):514-9. doi: 10.3345/kjp.2014.57.12.514. Epub 2014 Dec 31. PMID 25653684
- [Background] Nickeleit V, Hirsch HH, Zeiler M, Gudat F, Prince O, Thiel G, Mihatsch MJ. BK-virus nephropathy in renal transplants-tubular necrosis, MHC-class II expression and rejection in a puzzling game. Nephrol Dial Transplant. 2000 Mar;15(3):324-32. doi: 10.1093/ndt/15.3.324. PMID 10692517
- [Background] Cekmen MB, Bakirdoven S, Sayan M, Yilmaz A. BK virus nephropathy developing after renal transplantation and its treatment with ciprofloxacin: a case report. Transplant Proc. 2012 Dec;44(10):3044-7. doi: 10.1016/j.transproceed.2012.03.059. PMID 23195024
- [Background] Chalasani G, Li Q, Konieczny BT, Smith-Diggs L, Wrobel B, Dai Z, Perkins DL, Baddoura FK, Lakkis FG. The allograft defines the type of rejection (acute versus chronic) in the face of an established effector immune response. J Immunol. 2004 Jun 15;172(12):7813-20. doi: 10.4049/jimmunol.172.12.7813. PMID 15187165
- [Background] Zaman RA, Ettenger RB, Cheam H, Malekzadeh MH, Tsai EW. A novel treatment regimen for BK viremia. Transplantation. 2014 Jun 15;97(11):1166-71. doi: 10.1097/01.TP.0000441825.72639.4f. PMID 24531848
- [Background] Hoppe-Seyler K, Sauer P, Lohrey C, Hoppe-Seyler F. The inhibitors of nucleotide biosynthesis leflunomide, FK778, and mycophenolic acid activate hepatitis B virus replication in vitro. Hepatology. 2012 Jul;56(1):9-16. doi: 10.1002/hep.25602. Epub 2012 Jun 1. PMID 22271223
- [Background] Aldred KJ, Kerns RJ, Osheroff N. Mechanism of quinolone action and resistance. Biochemistry. 2014 Mar 18;53(10):1565-74. doi: 10.1021/bi5000564. Epub 2014 Mar 7. PMID 24576155
- [Background] Mateo R, Cho Y, Singh G, Stapfer M, Donovan J, Kahn J, Fong TL, Sher L, Jabbour N, Aswad S, Selby RR, Genyk Y. Risk factors for graft survival after liver transplantation from donation after cardiac death donors: an analysis of OPTN/UNOS data. Am J Transplant. 2006 Apr;6(4):791-6. doi: 10.1111/j.1600-6143.2006.01243.x. PMID 16539637
- [Background] Matsuoka L, Shah T, Aswad S, Bunnapradist S, Cho Y, Mendez RG, Mendez R, Selby R. Pulsatile perfusion reduces the incidence of delayed graft function in expanded criteria donor kidney transplantation. Am J Transplant. 2006 Jun;6(6):1473-8. doi: 10.1111/j.1600-6143.2006.01323.x. PMID 16686773
- [Background] Johnston TD, Thacker LR, Jeon H, Lucas BA, Ranjan D. Sensitivity of expanded-criteria donor kidneys to cold ischaemia time. Clin Transplant. 2004;18 Suppl 12:28-32. doi: 10.1111/j.1399-0012.2004.00214.x. PMID 15217404
- [Background] Israni AK, Salkowski N, Gustafson S, Snyder JJ, Friedewald JJ, Formica RN, Wang X, Shteyn E, Cherikh W, Stewart D, Samana CJ, Chung A, Hart A, Kasiske BL. New national allocation policy for deceased donor kidneys in the United States and possible effect on patient outcomes. J Am Soc Nephrol. 2014 Aug;25(8):1842-8. doi: 10.1681/ASN.2013070784. Epub 2014 May 15. PMID 24833128
- [Background] Duan KI, Englesbe MJ, Volk ML. Centers for Disease Control 'high-risk' donors and kidney utilization. Am J Transplant. 2010 Feb;10(2):416-20. doi: 10.1111/j.1600-6143.2009.02931.x. Epub 2009 Dec 2. PMID 19958324